CLINICAL TRIAL: NCT06870162
Title: Pain Disengagement Training: A Self-directed Intervention for Pain Catastrophizing (Open Pilot)
Brief Title: Pain Disengagement Training (Open Pilot)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Katherine A McDermott, Staff psychologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025p000348; 1K23AT012789-01 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-03

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: pain catastrophizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Disengagement Training (Experimental): The intervention involves approximately 8 sessions. The first session will involve a psychoeducation component describing the association between negative emotions and pain and the rationale for the intervention strategies. The intervention sessions will consist of approximately 30 minutes of writing alternating between imaginal exposure writing and positive writing periods alternating back and forth (e.g., 3-5 minutes of imaginal exposure writing followed by 3-5 minutes of positive writing before returning to imaginal exposure writing, etc.). Exposure writing will involve writing about a pain-related catastrophic worry repeatedly until it becomes less anxiety-provoking. The positive writing topics will change with each prompt and will be structured by session theme (e.g., values/goals, meaningful activities). They will also complete between session practice by setting aside a time for worrying and then completing a meaningful activity.
  Interventions: Behavioral: Pain Disengagement Training

INTERVENTIONS:
Behavioral: Pain Disengagement Training — The intervention involves approximately 8 sessions. The first session will involve a psychoeducation component describing the association between negative emotions and pain and the rationale for the intervention strategies. The intervention sessions will consist of approximately 30 minutes of writing alternating between imaginal exposure writing and positive writing periods alternating back and forth (e.g., 3-5 minutes of imaginal exposure writing followed by 3-5 minutes of positive writing before returning to imaginal exposure writing, etc.). Exposure writing will involve writing about a pain-related catastrophic worry repeatedly until it becomes less anxiety-provoking. The positive writing topics will change with each prompt and will be structured by session theme (e.g., values/goals, meaningful activities). They will also complete between session practice by setting aside a time for worrying and then completing a meaningful activity.

SUMMARY:
The investigators aim to conduct an open pilot trial to determine the initial feasibility of a self-directed writing-based intervention in individuals with chronic musculoskeletal pain and elevated pain catastrophizing. The investigators will assess the feasibility of recruitment, acceptability of the treatment, credibility and participant satisfaction, treatment adherence, and feasibility of assessments following pre-specified benchmarks.

DETAILED DESCRIPTION:
Mind-body interventions are some of the most effective treatments for chronic pain, yet due to lack of resources, many are inaccessible to the patients who need them. The investigators seek to fill this gap by developing and testing Pain Disengagement Training (PDT) for the treatment of chronic pain catastrophizing, a key risk factor for pain interference. The investigators will administer the PDT treatment in a small number (approximately 10) of participants to evaluate initial benchmarks (the feasibility of recruitment, acceptability of the treatment, credibility and participant satisfaction, treatment adherence, and feasibility of assessments) and to assess participants' experience with the intervention using qualitative exit interviews. Results will inform the refinement of the intervention for a future larger trial.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient adults (i.e., greater than or equal to 18)
2. Has self reported chronic musculoskeletal pain (i.e., pain persisting for at least 3 months)
3. Pain score greater than or equal to 4 (moderate) on the Numerical Rating Scale
4. Pain catastrophizing score greater than or equal to 20 on Pain Catastrophizing Scale
5. Willingness to engage in a writing-based intervention and self-reported ability to write or type for at least 30 minutes in a sitting
6. Received care at Massachusetts General Hospital
7. English verbal and writing fluency

Exclusion Criteria:

1. Clinically significant change in therapy or medication in the past 3 months
2. Severe untreated mental health condition (e.g., psychosis)
3. Active suicidality with history of plan or current intent
4. Serious illness expected to worsen in the next 6 months (e.g., cancer)
5. Untreated substance use problem that, per patient's self-report, would interfere with the ability to complete the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline, post-test (6 weeks)
  >70% participants approached agree to participate in the intervention
Acceptability of treatment | Baseline, post-test (6 weeks)
  >70% of participants attend at least 6 out of 8 sessions
Credibility and Expectancy Questionnaire | Baseline
  Measures perception that the treatment is credible and will offer improvements. Credibility (4 items) is rated from 1-9 with higher scores indicating more credibility. Expectancy is rated from 0-10 with higher scores indicating greater expectancy of improvement.
Client Satisfaction Questionnaire | Post-test (6 weeks)
  Measure of client satisfaction with a program or intervention. 8-item scale measured from 1 to 4 with greater scores indicating greater satisfaction.
Adherence to intervention | Mid-intervention
  Percent of writing sections demonstrate correct themes (e.g., anxiety words in imaginal exposure writing)
Feasibility of assessments | Baseline, post-test (6 weeks)
  >70% of participants have no measures fully missing

SECONDARY OUTCOMES:
Numerical Rating Scale | Baseline, post-test (6 weeks)
  Rating of pain intensity on a 0-10 1-item scale with greater scores indicating greater pain intensity
Graded Chronic Pain Scale | Baseline, post-test (6 weeks)
  Measure of pain severity. 3-item scale rated from 0 to 10 with greater scores indicating greater pain severity and interference
PROMIS Pain Interference scale | Baseline, post-test (6 weeks)
  Assesses pain interference in the past 7 days in activities, work, chores, etc. 8-item scale (1 - not at all to 5 - very much) with greater scores indicating greater pain interference.
Brief Pain Inventory | Baseline, post-test (6 weeks)
  Assesses pain intensity (4 items) on a 0 to 10 scale with greater scores indicating worse pain intensity and interference.
Patient Health Questionnaire - 9 | Baseline, post-test (6 weeks)
  Measure of depressive symptoms. 9-item scale rated from 0 to 3 with greater scores indicating greater depressive symptoms.
PROMIS depression scale-8 | Baseline, post-test (6 weeks)
  Measure of depressive symptoms. 8-item scale rated from 1 to 5 with greater scores indicating greater depressive symptoms.
Penn State Worry Questionnaire - abbreviated | Baseline, post-test (6 weeks)
  8-item measure of worry rated from 1 to 5 with greater scores indicating greater worry.
Pain Catastrophizing Scale | Baseline, post-test (6 weeks)
  Assesses magnification, helplessness, and rumination in response to pain. 13-item scale rated 0 to 4 with greater scores indicating greater pain catastrophizing.
Pain Anxiety Symptom Scale - Short Form (PASS-20) | Baseline, post-test (6 weeks)
  Assesses fear and anxiety in response to pain. 20-item scale rated 0 to 5 with greater scores indicating greater pain anxiety.
Worry Disengagement Questionnaire | Baseline, post-test (6 weeks)
  Measures ability to shift attention from worry. 4-item scale rated from 0 to 10 with greater scores indicating greater ability to shift attention away from worry.
Behavioral Activation for Depression Scale - Short Form | Baseline, post-test (6 weeks)
  Assesses engagement in meaningful activities. 9-item measure rated from 0 to 6 with greater scores indicating greater activity engagement.
Positive emotion rating scale | Mid-intervention
  Assesses level of emotional intensity on a 4-item scale from 1 to 5 with greater scores indicating more positive emotionality.
Contrast Avoidance Questionnaire-General Emotion and Worry subscales | Baseline, post-test (6 weeks)
  Measures ability to sustain negative emotionality to protect against sudden shifts in emotion. 25-item scale rated from 1 to 5 with greater scores indicating greater avoidance of contrasting emotional states.
PROMIS meaning and purpose scale short form 4a | Baseline, post-test (6-weeks)
  4 item scale assessing meaning and fulfillment in life (1 to 5 rating scale)
Self-Compassion Scale | Baseline, Post-test (6 weeks)
  12 item 1 to 5 scale measuring self-compassion

CONTACTS AND LOCATIONS:
Overall Officials: Katherine McDermott, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will include feasibility assessments, intervention measures (i.e., peak emotion during writing periods) and pre and post intervention self-report questionnaires in the open pilot.
Supporting Information: SAP, Analytic Code
Time Frame: Data from this study will be deposited into the repositories no later than the end of the funded project period. Data will be available indefinitely and will only be removed from the repository if requested by NIH or other relevant institution policy.
Access Criteria: Data will be stored in the Vivli repository, an NIH-approved independent, generalist global data-sharing and analytics platform. Researchers will be able to access the data by request. Investigators will need to provide evidence of their institution's IRB approval for planned analyses of the data and upon the contingency that data only be used for research and secured by electronic safeguards. Further, this agreement will state that data will be destroyed once data analysis is complete.
URL: https://vivli.org/